CLINICAL TRIAL: NCT06072261
Title: The Effect of Handgrip Strength on Functional Level in Elderly People Having Lower Extremity Surgery
Brief Title: The Effect of Handgrip Strength on Functional Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Menekse Safak, Research Assistant, Suleyman Demirel University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MS2023/02
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Rehabilitation
Keywords: Elderly; Functional Level; Handgrip Strenght; Kinesio Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Tape Group (Experimental): Before the standard rehabilitation program, kinesio taping was applied to both upper extremities in the form of a "Y" tape from the medial epicondyle to the wrist flexors, with 15-20% tension, to the patients hospitalized in the orthopedic service after lower extremity surgery. The tape should remain on the patient's arm throughout the hospital stay
  Interventions: Other: kinesio tape application
- Control Group (No Intervention): For the control group data, patients who underwent lower extremity surgery at the same institution for similar periods, but were included in the standard rehabilitation program, but did not apply kinesio tape, will be included. Standard rehabilitation practice includes in-bed transfer training, gait training, practice of daily living activities, and therapeutic exercise practices

INTERVENTIONS:
Other: kinesio tape application — Before the standard rehabilitation program, kinesio taping was applied to both upper extremities in the form of a "Y" tape from the medial epicondyle to the wrist flexors, with 15-20% tension, to the patients hospitalized in the orthopedic service after lower extremity surgery. The tape should remain on the patient's arm throughout the hospital stay
  Arms: Kinesio Tape Group

SUMMARY:
In this study, it was aimed to examine the effects of kinesio tape applied to the forearm extensor muscles on the functional level of patients undergoing lower extremity surgery with walker ambulation.

Patients who were evaluated before being included in the post-surgical rehabilitation program (before kinesio tape application) and before discharge will be included in the study group. For the control group data, patients who underwent lower extremity surgery at the same institution for similar periods, but were included in the standard rehabilitation program, but did not apply kinesio tape, will be included. Standard rehabilitation practice includes in-bed transfer training, gait training, practice of daily living activities, and therapeutic exercise practices .

Before the standard rehabilitation program, kinesio taping was applied to both upper extremities in the form of a "Y" tape from the medial epicondyle to the wrist flexors, with 15-20% tension, to the patients hospitalized in the orthopedic service after lower extremity surgery. The tape should remain on the patient's arm throughout the hospital stay

DETAILED DESCRIPTION:
In the literature, as predictors of poor functional recovery after lower extremity fracture and prosthetic surgery; old age, low functional level before fracture, cognitive impairment, comorbidities, living alone, and long hospital stay have been shown. Although the lower extremity has a higher relationship than the upper extremity in activities such as walking and physical function, the grip strength, which is closely related to the lower extremity strength, is an easily measurable, reliable, and applicable method for assessing whole body strength.In addition, handgrip strength is used as an important criterion in determining the functional level of elderly individuals. Although there are many studies in the literature that grip strength is a determinant of functional level, no study has been encountered showing the effects of kinesio taping application on the functional level of improving grip strength in elderly individuals who have undergone lower extremity surgery and provided with walker assisted ambulation.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 65 years of age of both sexes, patients who were followed up postoperatively in the Department of Orthopedics of Süleyman Demirel University, patients whose mobilization was provided with a walker, and patients whose general condition was oriented and cooperative, were included in the study

Exclusion Criteria:

* Patients with uncontrollable lung or cardiac problems, patients with psychiatric disease (dementia…) that may affect the answers given, patients who used any drugs and alcohol that could affect cognitive functions were excluded from the study.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Handgrip strenght | 3-5 days (Change from Baseline Handgrip strenght at discharged)
  It was evaluated using a Jamar handheld dynamometer. During the evaluation, the patient was asked to stand in a static position. Maximum grip strength measurements were performed with the elbow flexed at 90° in the patient sitting position. Measurements were repeated 3 times at 30 second intervals in both extremities, and the results were recorded in kilogram-force form. In the measurement of maximum handgrip strength, the participants were asked to continue squeezing even if there was pain, and the maximum grip strength they reach was recorded
Pain assessment | 3-5 days (Change from Baseline Handgrip strenght at discharged)
  Visual Analogue Scale (VAS) was used for pain assessment. The pain of the patient, who determines a point on the vertically drawn line with a length of 10 cm, is determined over one hundred points. A score of 100 means unbearable pain, and a score of 0 means no pain at all. This evaluation provides information about the pain profile of patients during activity and at rest
Functional Independence Measurement-FIM | 3-5 days (Change from Baseline Handgrip strenght at discharged)
  The FIM instrument FIM indicates the degree of independence of the individual in basic physical and cognitive activities in daily life. The FIM includes 18 items that measure functional independence in 6 subscales: self-care, sphincter control, mobility, locomotion, communication, and social cognition. Each item is rated on a seven-point scale that represents different gradations of independence and reflects the amount of assistance the patient requires to perform a specific activity. Independence is categorized and scored as complete independence, 7; modified independence, 6; requires supervision or setup, 5; requires minimal contact assistance, 4; requires moderate assistance, 3; requires maximal assistance, 2; and requires total assistance, 1. The sum of all 18 items comprises the patient's total FIM score, which ranges from 18 to 126
Iowa Level of Assistance Scale (ILAS) and Walking Speed Scale (IWSS) | 3-5 days (Change from Baseline Handgrip strenght at discharged)
  ILAS and IWSS are a measurement method that evaluates various physical functions and whose validity and reliability have been demonstrated in patients with knee replacement. With the ILAS, the performance level of 4 different physical activities (from lying on the back to sitting, getting up from sitting, walking 4.57 meters (15 feet), going up and down three flights of stairs) is evaluated. The scoring of these physical activities is based on the level of assistance that patients need during the activities ("0" could not be tested, "1" unsuccessful, "2" maximum assistance, "3" medium assistance, "4" minimum assistance, "5" observational assistance, "5" observational assistance. 6" independent) are made. With IWSS, walking speed is evaluated at a distance of 13.4 meters (44 feet). This scale ranges from 0 to 6 ("0" ≤20 sec, "1" 21-30 sec, "2" 31-40 sec, "3" 41-50 sec, "4" 51-60 sec, "5" 61 -70 sec, "6" >70 sec) or the time to complete walking is recorded as a score.

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha BAŞKURT, Prof. Dr., Principal Investigator — Suleyman Demirel University; Ferdi BAŞKURT, Prof. Dr., Study Chair — Suleyman Demirel University; Tuba İNCE PARPUCU, Assist. Prof., Study Chair — Suleyman Demirel University
Locations (1):
- Menekşe ŞAFAK, Merkez, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No